CLINICAL TRIAL: NCT00233038
Title: EUS-Guided Pancreatic Injection of Cyst (EPIC) Trial
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Indiana University School of Medicine (Other)
Responsible Party: Principal Investigator, William R. Brugge, MD, Director of Pancreas and Biliary Center, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2003-P-001745
Record Dates: First submitted 2005-10-03; First posted 2005-10-05 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-10

CONDITIONS: Pancreatic Cystadenoma
Keywords: Pancreatic cancer; Pancreatic adenoma; Ethanol; Endoscopic ultrasound; Cyst ablation
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatic adenoma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Ethanol injection into a cyst

SUMMARY:
The purpose of the study is to learn about a new treatment for pancreatic cystic lesions. The injection of alcohol into cysts is a common way of treating cysts of the liver, kidney, and thyroid. We would like to find out if injection of alcohol would be useful for the treatment of pancreatic cystic lesions. The treatment with alcohol will use endoscopy and endoscopic ultrasound (procedures that use a scope that is placed through your mouth and into your stomach). We hypothesize that more than half of the cysts which are injected with ethanol will resolve.

DETAILED DESCRIPTION:
Cystic lesions of the kidney, thyroid, and liver are commonly treated with ethanol injections into the cyst cavity. The contact with ethanol results in rapid elimination of epithelial cells lining cyst cavities with few complications or pain. The majority of cysts become smaller and some are completely eliminated Depending on the type of cyst and tissue, some cysts can be completely ablated with ethanol. Although malignant masses arising from the pancreas have been safely injected with ethanol, there are no reports of injection of pancreatic cystadenomas. The ability to ablate cystadenomas of the pancreas would provide the first non-surgical treatment for these pre-malignant lesions of the pancreas.

Over the past two years we have conducted a pilot study of EUS-guided ethanol lavage of pancreatic cysts (2001-P-000358/5). 18 patients have undergone the procedure without evidence of pancreatitis, pain, or infection following the procedure. Initially, low concentrations of ethanol were used (5%) and over the course of the study, the concentration of the ethanol used for lavage has been increased to 60%. Although the patients have not undergone careful follow-up evaluations, it appears that at least 4 of the patients have had resolution of the cyst.

This is a prospective, randomized, blinded, controlled trial of ethanol ablation in 50 patients with a pancreatic cystadenoma. Patients with a pancreatic cyst (1-5cm in diameter) capable of safely undergoing endoscopy with conscious sedation will be candidates. Exclusion criteria include: coagulopathy (INR>1.5, PTT>100, platelets of< 50k), active infection of the cyst or unstable cardio-pulmonary disease (active angina, home O2, or pulmonary edema) will be excluded.

At the time of diagnostic cyst aspiration, the patient will be randomized to either saline lavage or ethanol (70%) lavage. During the exam, the cyst will be imaged with ultrasound, measured and aspirated. The cyst contents will be evaluated with cytologic evaluation, CEA, and amylase. After cyst aspiration, the cyst will be lavaged with either saline or ethanol for 5 minutes. At completion of the lavage, the cyst contents will be evacuated. The patient will be provided the results of the cyst fluid analysis and may elect to undergo surgical resection or additional lavage treatments. At the time of resection, the cyst and surrounding pancreas will be resected for histologic analysis. The degree of epithelial ablation will be determined with histologic sectioning and the cysts lavaged with ethanol will be compared to those cysts lavaged with saline. If the patient chooses not to have a surgical resection, the patient may return for a follow-up EUS exam at two additional monthly intervals with cyst aspiration and additional ethanol lavage. Those patients receiving saline during the initial treatment session will be crossed-over to ethanol.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a pancreatic cyst (1-5cm in diameter)
* Capable of safely undergoing endoscopy with conscious sedation

Exclusion Criteria:

* Coagulopathy (INR>1.5, PTT>100, platelets of< 50k)
* Active infection of the cyst
* Unstable cardio-pulmonary disease (active angina, home O2, or pulmonary edema)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-01; Primary Completion 2007-12 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William R. Brugge, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Indiana University Medical Center, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Kim KH, McGreevy K, La Fortune K, Cramer H, DeWitt J. Sonographic and cyst fluid cytologic changes after EUS-guided pancreatic cyst ablation. Gastrointest Endosc. 2017 Jun;85(6):1233-1242. doi: 10.1016/j.gie.2016.09.011. Epub 2016 Sep 17. PMID 27650271
- [Derived] DeWitt J, McGreevy K, Schmidt CM, Brugge WR. EUS-guided ethanol versus saline solution lavage for pancreatic cysts: a randomized, double-blind study. Gastrointest Endosc. 2009 Oct;70(4):710-23. doi: 10.1016/j.gie.2009.03.1173. Epub 2009 Jul 4. PMID 19577745